CLINICAL TRIAL: NCT02417831
Title: Single Center, Single Dose, Open-label, Randomized, Two-way Crossover Study to Determine Bioequivalence of Two Formulations Containing Tamsulosin HCl 04.mg MR Capsules in at Least 30 Healthy Male Subjects Under Fasted Conditions
Brief Title: Determine the Bioequivalence of Two Formulations of Tamsulosin HCl Capsules in Fasted Male.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 527.88
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

ARMS (2):
- tamsulosin capsules (Active Comparator)
  Interventions: Drug: tamsulosin capsules
- tamsulosin HCl capsules (Active Comparator)
  Interventions: Drug: tamsulosin HCl

INTERVENTIONS:
Drug: tamsulosin capsules
  Arms: tamsulosin capsules
Drug: tamsulosin HCl
  Arms: tamsulosin HCl capsules

SUMMARY:
A bio-equivalence of 2 different capsule formulations in fasted subjects

ELIGIBILITY:
Inclusion criteria:

Healthy male volunteers 18 years and older

Exclusion criteria:

History of hypersensitivity or allergy to the IPM or its excipients or any related medication

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Groups:
- New MR (Test) / Registered MR (Reference): Oral administration of tamsulosin new 0.4mg modified release (MR) capsule followed by oral administration of tamsulosin registered 0.4mg MR capsule in the fasted state after an overnight fast of at least 10 hours. Treatment periods were separated by a wash-out period of 07 days.
- Registered MR (Reference) / New MR (Test): Oral administration of tamsulosin registered 0.4mg MR capsule followed by oral administration of tamsulosin new 0.4mg MR capsule in the fasted state after an overnight fast of at least 10 hours. Treatment periods were separated by a wash-out period of 07 days.
Period: Period 1: Treatment Period 1 + Washout
Arm/Group | New MR (Test) / Registered MR (Reference) | Registered MR (Reference) / New MR (Test)
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Period 2: Treatment Period 2 + Washout
Arm/Group | New MR (Test) / Registered MR (Reference) | Registered MR (Reference) / New MR (Test)
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who received at least one dose of investigational medicinal product.
Groups:
- All Subjects: Subjects each received two treatments which were each administered orally in the fasted state after an overnight fast of at least 10 hours. and separated by a washout period of 7 days. The treatments were:
  * New MR (Test): Tamsulosin 0.4mg modified release (MR) capsule.
  * Registered MR (Reference) : Tamsulosin 0.4mg capsule.
Arm/Group | All Subjects
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum measured concentration in plasma (Cmax). Geometric Coefficient of Variation (gCV) is actually inter-individual gCV.
Time Frame: Before drug administration (0 hours (h)) and 1h, 2h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h and 72h after drug administration.
Population: Pharmacokinetic set (PK set): All subjects who had evaluable pharmacokinetic (PK) data for both treatment periods were included in the statistical PK analysis for the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- New MR (Test): Oral administration of tamsulosin new 0.4mg modified release (MR) capsule.
- Registered MR (Reference): Oral administration of tamsulosin registered 0.4mg MR capsule.
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
pg/mL | 21700 (37.8) | 20520 (36.7)
Statistical Analysis 1: Comparison: New MR (Test) vs Registered MR (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Ratio = 105.76, 90% CI 2-sided [99.81 to 112.08], Standard Deviation 14.18 — The standard deviation in the statistical analysis is actually the intra-individual coefficient of variation. Ratio calculated as test divided by reference

2. Primary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz).
  Geometric Coefficient of Variation (gCV) is actually inter-individual gCV.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
h*pg/mL | 241500 (48.4) | 238200 (48.0)
Statistical Analysis 1: Comparison: New MR (Test) vs Registered MR (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Ratio = 101.40, 90% CI 2-sided [97.71 to 105.23], Standard Deviation 9.05 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: (AUC0-inf)
Description: Area under the concentration-time curve of analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
  Geometric Coefficient of Variation (gCV) is actually inter-individual gCV.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
h*pg/mL | 248200 (49.4) | 244700 (48.9)
Statistical Analysis 1: Comparison: New MR (Test) vs Registered MR (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Ratio = 101.42, 90% CI 2-sided [97.81 to 105.17], Standard Deviation 8.85 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Tmax
Description: Time to maximum plasma concentration
Time Frame: as for outcome 1
Population: PK set
Measure: Median (Full Range); unit: Hours
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
Hours | 5.004 [3.00 to 6.00] | 5.006 [3.00 to 8.01]

5. Secondary Outcome: λz
Description: Terminal elimination rate constant in plasma (λz).
  Geometric Coefficient of Variation (gCV) is actually inter-individual gCV.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hours
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
1/hours | 0.05 (28.40) [0.0338 to 0.133] | 0.05 (24.10) [0.0347 to 0.0766]

6. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life of the analyte in plasma (t1/2)
  Geometric Coefficient of Variation (gCV) is actually inter-individual gCV.
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | New MR (Test) | Registered MR (Reference)
Number analyzed (Participants) | 34 | 34
Hours | 13.10 (28.40) [5.22 to 20.5] | 13.52 (24.10) [9.04 to 20.0]

ADVERSE EVENTS:
Time Frame: From drug administration until 7days thereafter for each treatment arm, upto 10 days.
Arm/Group | New MR (Test) | Registered MR (Reference)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 6/34 | 9/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New MR (Test) (N=34) | Registered MR (Reference) (N=34)
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.